CLINICAL TRIAL: NCT06851195
Title: Effect of Neuromuscular Electrical Stimulation of Lower Limbs on Improving Exercise Self-Efficacy, Dyspnea During Activity and Fatigue in Patients With Chronic Obstructive Pulmonary Disease
Acronym: NMES
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KMUHIRB-F(II)-20240343
Record Dates: First submitted 2025-02-20; First posted 2025-02-28 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-01

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD); Neuromuscular Electrical Stimulation (NMES); Exercise Self-Efficacy; Dyspnea During Activity; Fatigue
Keywords: Chronic Obstructive Pulmonary Disease (COPD); Neuromuscular Electrical Stimulation (NMES); Exercise Self-Efficacy; Dyspnea During Activity; Fatigue
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- neuromuscular electrical stimulation (Experimental): lower limb neuromuscular electrical stimulation
- routine treatment：Pulmonary rehabilitation exercises (Other): The control group only participated in the lung rehabilitation exercise program (after which the control group received electrical stimulation for two months)
  Interventions: Behavioral: pulmonary rehabilitation exercises

INTERVENTIONS:
Device: lower limb neuromuscular electrical stimulation — The study adopts a quasi-experimental design with convenience sampling. Data collection will be done through structured questionnaires. Patients who meet the inclusion criteria will be referred by physicians, and before enrollment, a verbal introduction will be given explaining the study's purpose, the questionnaire, and the intervention procedure and duration. The experimental group will participate in both pulmonary rehabilitation exercises and an additional intervention of lower limb neuromuscular electrical stimulation, 30 minutes per session, three times per week, for eight weeks. The control group will only participate in pulmonary rehabilitation exercises. Based on Hill et al. (2018), neuromuscular electrical stimulation should continue for 4 to 8 weeks. Questionnaires will be administered before the intervention and at the 2nd, 4th, 6th, and 8th weeks post-intervention, including basic information, Modified Medical Research Council Dyspnea Scale, Manchester COPD Fatigue Scale,
Behavioral: pulmonary rehabilitation exercises — The control group only participated in the lung rehabilitation exercise program (after which the control group received electrical stimulation for two months)
  Arms: routine treatment：Pulmonary rehabilitation exercises

SUMMARY:
Patients diagnosed with COPD who meet the inclusion and exclusion criteria, either inpatients or outpatients, will be informed about the study'sstudy's purpose and procedures by the principal investigator. After understanding their rights, they will provide informed consent.

DETAILED DESCRIPTION:
The process of the experiment The study adopts a quasi-experimental design with convenience sampling. Data collection will be done through structured questionnaires. Patients who meet the inclusion criteria will be referred by physicians, and before enrollment, a verbal introduction will be given explaining the study's purpose, the questionnaire, and the intervention procedure and duration. The experimental group will participate in both pulmonary rehabilitation exercises and an additional intervention of lower limb neuromuscular electrical stimulation, 30 minutes per session, three times per week, for eight weeks. The control group will only participate in pulmonary rehabilitation exercises. Neuromuscular electrical stimulation should continue for 4 to 8 weeks. Questionnaires will be administered before the intervention and at the 2nd, 4th, 6th, and 8th weeks post-intervention, including basic information, Modified Medical Research Council Dyspnea Scale, Manchester COPD Fatigue Scale, and Self-Efficacy for Exercise Scale. Data collection will take approximately 25 minutes, and questionnaires will be personally retrieved by the researcher.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with COPD as per pulmonary function reports, with post-bronchodilator FEV1/FVC ratio < 0.7, confirmed as mild to severe COPD by physician, without acute exacerbation, aged 18 or above, enrolled in a pulmonary rehabilitation program, able to communicate clearly in Mandarin or Taiwanese, and without history of a psychiatric disorders.

Exclusion Criteria:

* Patients unable to comply with long-term follow-up for lower limb neuromuscular electrical stimulation intervention, those with cardiac pacemakers, lower limb bone, joint, or neuromuscular diseases, obesity (BMI >35 kg/m2), or systemic vascular diseases (e.g., lupus erythematosus).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change exercise self-efficacy | 8 weeks
  This scale is used to assess an individual's confidence in performing exercise behaviors when faced with various situations that are not conducive to exercise. The Chinese version of the Sports Self-efficacy Scale consists of 10 questions, scored from 0 to 10, to understand the degree of confidence in engaging in sports. "0" represents little confidence, and "10" represents great confidence. The higher the score, the more confident one is in performing sports in the face of various situations and obstacles.
change dyspnea during activity | 8 weeks
  Modified Medical Research Council(mMRC)
change fatigue | 8 weeks
  The Manchester fatigue scale (MFS) is divided into three aspects, including fatigue conditions such as physiological level (11 questions), cognitive feelings (9 questions) and psychosocial function (7 questions). There are 27 questions in total, with a five-point scoring method. The scoring method is 1 point for "never", 2 points for "rarely", 3 points for "sometimes", 4 points for "often", and 5 points for "always". The higher the score, the higher the degree of fatigue.

SECONDARY OUTCOMES:
Short Physical Performance Battery | 8 weeks
  The project leader will collect data on the Short Physical Performance Battery (SPPB) before the intervention and eight weeks after the intervention. If there is no pre-test data of the Short Physical Performance Battery (SPPB), the Short Physical Performance Battery (SPPB) will be administered again two months after the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No